CLINICAL TRIAL: NCT05378321
Title: The Prevalence of Non-Alcoholic Fatty Liver Disease in Patients With an Acute Cardiac Event Followed at Ziekenhuis Oost-Limburg, Genk, Belgium
Brief Title: Prevalence of NAFLD in ACS Patients
Acronym: PADAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Mathieu Struyve, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PADAC-01
Record Dates: First submitted 2022-04-13; First posted 2022-05-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: NAFLD; ACS - Acute Coronary Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ACS risk gropu (Other): Group of patients with an acute-cardiovascular syndrome.
  Interventions: Diagnostic Test: Non-invasive diagnostic testing

INTERVENTIONS:
Diagnostic Test: Non-invasive diagnostic testing — Non-invasive diagnostic testing consists of the use of the FibroScan device and the calculation of non-invasive blood-based scores for the diagnosis of NAFLD

SUMMARY:
Addressing CVD risk in patients with NAFLD is the aspect of the disease most amenable to medical management and so improving long-term clinical outcomes. Almost no studies have been done concerning the prevalence of NAFLD in CVD patients, most of the conducted studies have been done in already diagnosed NAFLD patients to estimate the risk of CVD development. Currently, there are no data available about the prevalence of NAFLD in CVD, more specifically patients with an acute cardiovascular event (ACE) in Belgium.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* having acute cardiovascular syndrome
* able to understand Dutch
* able to understand the informed consent

Exclusion Criteria:

* excessive alcohol abuse
* other liver disease
* secondary causes of steatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
FibroScan® liver stiffness measurements | 4 years
  The FibroScan® device measures vibration controlled transient elastography (VCTE) (kPa) Based on these values the liver stiffness status will be determined.
FibroScan® steatosis measurements | 4 years
  The FibroScan® device measures controlled attenuation parameter (CAP) (dB/m) Based on these values the liver steatosis status will be determined.
Liver ultrasound | 4 years
  Out of the EPF the results of a possible earlier ultrasound are noted in the CRF. The results are noted as 'liver steatosis found' with yes/no answer and the year in which this ultrasound was performed.
Liver biopsy results | 4 years
  Out of the EPF the results of a possible earlier ultrasound or liver biopsy are noted in the CRF. The NAS CRN (histological) score is noted. The score ranges from 0-8 and is composed of the unweighted sum of steatosis, ballooning, and lobular inflammation. A score between 0-2 corresponds to no NASH, 3-4 is borderline NASH, and definite NASH has a score between 5 and 8.
Aspartate transaminase (AST) | 4 years
  Out of the EPF the blood parameter AST (U/L) will be collected.
Alanine transaminase (ALT) | 4 years
  Out of the EPF the blood parameter ALT (U/L) will be collected.
Gamma glutamyltransferase (GGT) | 4 years
  Out of the EPF the blood parameter GGT (U/L) will be collected.
Lactate dehydrogenase (LDH) | 4 years
  Out of the EPF the blood parameter LDH (U/L) will be collected.
Exclusion of other liver diseases | 4 years
  hepatitis B, hepatitis C, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson disease and alpha 1 antitrypsin deficiency. NAFLD is a disease of exclusion and therefore the abovementioned parameters are determined out of the EPF.
Wellbeing - BAECKE | 4 years
  This questionnaire will be used to estimate the level of physical activity. It exists out of 16 questions about work, sports and leisure time. A higher score means that the person is more active at work, does more sport and has a more active leisure time. Minimum value is 3 and maximum value is 15.
Wellbeing - GAD-7 | 4 years
  General Anxiety Disorder (GAD-7) questionnaire will be used to determine the presence of possible clinically significant anxiety disorder. A higher scores indicates having anxiety. Minimum score is 0 and maximum score is 21.
Wellbeing - PHQ-9 | 4 years
  Patient Health Questionnaire-9 (PHQ-9) will be used to quantify depression symptoms and monitor severity. Minimum score is 0 and maximum score is 27. A higher score indicates having a depression.
Wellbeing - WPAI-SHP | 4 years
  Workers Productivity and Activity Impairment (WPAI-SHP) questionnaire. By means of 6 questions about work productivity and activity it can be determined if there is absence, productivity loss or a decrease in activities at work. The score is expressed in percentages (0-100). A higher percentage indicates a higher absence from work and a lower productivity.
Wellbeing-SF-36 | 4 years
  Short Form Health Survey-36 will be used to determine the health related quality of life based on 6 different topics: physical functioning, social functioning, role restrictions, mental wellbeing, energy and pain. The score is expressed in percentages (0-100). A higher percentage indicates a better general wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided